CLINICAL TRIAL: NCT04824833
Title: The Effects of Ultrasound-guided Serratus Anterior Plane Block on Intraoperative Opioid Consumption and Hemodynamic Stability During Breast Surgery: A Randomized Controlled Study
Brief Title: Effects of US-guided SAPB During Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Çağdaş Baytar, medical doctor, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2021/03-12
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Hemodynamic Instability; Opioid Use; Block; Breast Cancer
Keywords: hemodynamics; serratus anterior plane block; opioid consumption; breast surgery
MeSH Terms: conditions — Bites and Stings; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus anterior plane block (Active Comparator)
  Interventions: Procedure: Serratus anterior plane block
- control group (No Intervention)

INTERVENTIONS:
Procedure: Serratus anterior plane block — local anesthetic application between serratus anterior muscle and 5th rib
  Arms: Serratus anterior plane block

SUMMARY:
The serratus anterior plan (SAP) block is a technique that has recently gained popularity in the context of breast surgery. SAP block resulted in better hemodynamic stability, early ambulation and shorter hospital stay, as well as hospital costs for postoperative breast patients.

We aimed to investigate the effects of the serratus anterior plane block in women undergoing breast surgery, in the intraoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-75,
* ASA I-II-III risk group
* Patients who underwent breast surgery under general anesthesia, who underwent serratus anterior plan block for analgesia, or who were provided analgesia with conventional methods
* Patients whose informed consent was read and whose consent was obtained

Exclusion Criteria:

* who do not want to participate in the study,
* ASA IV-V patients

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
hemodynamic stability | during surgery
  effect of serratus anterior plane block on hemodynamic stability during breast surgery
opioid consumption | during surgery
  effect of serratus anterior plane block on opioid consumption during breast surgery

SECONDARY OUTCOMES:
emergence time | end of the surgery
  the time period between surgical incision closure and extubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University medicine faculty, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baytar C, Aktas B, Aydin BG, Piskin O, Cakmak GK, Ayoglu H. The effects of ultrasound-guided serratus anterior plane block on intraoperative opioid consumption and hemodynamic stability during breast surgery: A randomized controlled study. Medicine (Baltimore). 2022 Sep 2;101(35):e30290. doi: 10.1097/MD.0000000000030290. PMID 36107549